CLINICAL TRIAL: NCT01194245
Title: A Phase II, Randomized, Double Blind, 2-Way Crossover Safety and Efficacy Study of Subcutaneously Injected Prandial Insulins: Lispro-PH20 or Aspart-PH20 Compared to Insulin Lispro (Humalog®) in Patients With Type 1 Diabetes
Brief Title: Safety/Efficacy Study of Subcutaneously Injected Prandial Insulins Compared to Insulin Lispro Alone in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HALO-117-205
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart; insulin glulisine; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lispro-PH20 / Insulin Lispro (Experimental): All enrolled participants underwent a titration period of 4-6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually.
  Next participants were randomly assigned to 1 of 2 study treatments (Treatment A or B) for the first of two, 3-month treatment cycles. Each participant then received the second treatment for the second cycle with no washout period.
  Lispro-PH20 (Treatment A): 100 U/mL insulin lispro with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected SC, pre-meals, with doses titrated to each participant individually
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
  Interventions: Drug: Insulin lispro; Drug: recombinant human hyaluronidase PH20; Drug: Insulin glulisine; Drug: Insulin glargine
- Aspart-PH20 / Insulin Lispro (Experimental): All enrolled participants underwent a titration period of 4-6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually.
  Next participants were randomly assigned to 1 of 2 study treatments (Treatment A or B) for the first of two, 3-month treatment cycles. Each participant then received the second treatment for the second cycle with no washout period.
  Aspart-PH20 (Treatment A): 100 U/mL insulin aspart with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected SC, pre-meals, with doses titrated to each participant individually
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
  Interventions: Drug: Insulin lispro; Drug: recombinant human hyaluronidase PH20; Drug: Insulin aspart; Drug: Insulin glulisine; Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin lispro
  Other Names: Humalog
Drug: recombinant human hyaluronidase PH20
  Other Names: Hylenex; rHuPH20; PH20
Drug: Insulin aspart
  Arms: Aspart-PH20 / Insulin Lispro
Drug: Insulin glulisine
  Other Names: Apidra
Drug: Insulin glargine
  Other Names: Lantus

SUMMARY:
The purpose of the study is to compare Humalog (Insulin lispro)-recombinant human hyaluronidase (rHuPH20) or Novolog (Insulin aspart)-rHuPH20 to Humalog (Insulin lispro) for the treatment of Type 1 Diabetes Mellitus (T1DM) in basal-bolus therapy.

DETAILED DESCRIPTION:
Criteria for randomization into the study included 1) fasting blood glucose and predinner glucose values in the range of 70 to 140 milligrams per deciliter (mg/dL) approximately 60% of the time for 7 days prior to randomization 2) 90 minute or 2-hour postprandial blood glucose <220 mg/dL approximately 70% of the time for 7 days prior to randomization and 3) successfully completed 3 days of 10-point glucose monitoring and have at least 4 self-monitored blood glucose values on all non-10-point monitoring days. Participants that did not meet 1 or more of these criteria during a 4- to 6-week Titration Period were not randomized.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years
* Type 1 Diabetes Mellitus (T1DM) treated with insulin for ≥12 months
* Body mass index (BMI) 18.0 to 40.0 kilograms per square meter (kg/m^2).
* Hemoglobin A1C (HbA1C) level 6.7% to 8.2%, inclusive
* Fasting C-peptide <0.6 nanograms per milliliter (ng/mL)
* Willingness to use twice daily (BID) insulin glargine as basal insulin for the duration of the study
* Willingness to avoid use of an insulin infusion pump or unblinded continuous glucose monitoring (CGM) during the study

Exclusion Criteria:

* Known or suspected allergy to any component of any of the study drugs
* Use of pramlintide within 30 days of Screening
* Use of drugs during the study or within 30 days of Screening (such as corticosteroids or antimetabolites) that could interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia
* Recurrent severe hypoglycemia (more than 2 episodes over the last 6 months) or hypoglycemic unawareness, as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Muchmore, M.D., Study Director — Halozyme Therapeutics
Locations (19):
- United States (19):
  - AMCR Institute, Inc., Escondido, California
  - Scripps Whittier Diabetes Institute, La Jolla, California
  - Mills-Peninsula Health Services, San Mateo, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Diabetes Research Institute, Miami, Florida
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Mid-America Diabetes Associates, Wichita, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Medstar Research Institute, Hyattsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Mercury Street Medical, Butte, Montana
  - Desert Endocrinology, Henderson, Nevada
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Cetero Research-San Antonio, San Antonio, Texas
  - West Olympia Internal Medicine, Olympia, Washington
  - University of Washington School of Medicine, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included an open-label titration period of at least 4 weeks and up to 6 weeks prior to randomization at Week 0.
Groups:
- All Enrolled Participants: Prior to randomization, all enrolled participants underwent a titration period of 4-6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually.
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Lispro-PH20 First, Then Insulin Lispro: Following a titration period of 4 to 6 weeks, participants were randomly assigned to Treatment A for the first 3-month treatment cycle, followed by Treatment B for the second 3-month treatment cycle.
  Lispro-PH20 (Treatment A): 100 units per milliliter (U/mL) insulin lispro with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Insulin Lispro First, Then Lispro-PH20: Following a titration period of 4 to 6 weeks, participants were randomly assigned to Treatment B for the first 3-month treatment cycle, followed by Treatment A for the second 3-month treatment cycle.
  Insulin Lispro (Treatment B): 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Lispro-PH20 (Treatment A): 100 U/mL insulin lispro with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected SC, pre-meals, with doses titrated to each participant individually
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Aspart-PH20 First, Then Insulin Lispro: Following a titration period of 4 to 6 weeks, participants were randomly assigned to Treatment A for the first 3-month treatment cycle, followed by Treatment B for the second 3-month treatment cycle.
  Aspart-PH20 (Treatment A): 100 units per milliliter (U/mL) insulin aspart with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Insulin Lispro First, Then Aspart-PH20: Following a titration period of 4 to 6 weeks, participants were randomly assigned to Treatment B for the first 3-month treatment cycle, followed by Treatment A for the second 3-month treatment cycle.
  Insulin Lispro (Treatment B): 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Aspart-PH20 (Treatment A): 100 U/mL insulin aspart with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected SC, pre-meals, with doses titrated to each participant individually
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
Period: Titration Period (4 to 6 Weeks)
Arm/Group | All Enrolled Participants | Lispro-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Lispro-PH20 | Aspart-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Aspart-PH20
Started | 135 | 0 | 0 | 0 | 0
Completed | 117 (Participants that completed the Titration Period were randomized to Treatment Period 1.) | 0 | 0 | 0 | 0
Not Completed | 18 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0 | 0
Not completed — Titration Failure | 3 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Randomization Criteria | 7 | 0 | 0 | 0 | 0
Period: Treatment Period 1 (Weeks 0 to 12)
Arm/Group | All Enrolled Participants | Lispro-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Lispro-PH20 | Aspart-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Aspart-PH20
Started | 0 | 29 | 28 | 30 | 30
Received at Least 1 Dose of Study Drug | 0 | 29 | 28 | 30 | 30
Completed | 0 | 29 | 27 | 29 | 28
Not Completed | 0 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1
Period: Treatment Period 2 (Weeks 12 to 24)
Arm/Group | All Enrolled Participants | Lispro-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Lispro-PH20 | Aspart-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Aspart-PH20
Started | 0 | 29 | 27 | 29 | 28
Completed | 0 | 29 | 27 | 29 | 28
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Non-randomized Participants: Participants underwent a titration period of 4-6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually. Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
  Participants did not complete the titration period or did not meet one or more randomization criteria and, therefore, were not randomized.
- Total: Total of all reporting groups
Arm/Group | Non-randomized Participants | Lispro-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Lispro-PH20 | Aspart-PH20 First, Then Insulin Lispro | Insulin Lispro First, Then Aspart-PH20 | Total
Number analyzed (Participants) | 18 | 29 | 28 | 30 | 30 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (11.71) | 44.6 (14.56) | 45.7 (14.94) | 42.8 (14.13) | 42.5 (14.70) | 42.6 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 13 | 14 | 15 | 61
  Male | 12 | 16 | 15 | 16 | 15 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 2 | 3
  White | 17 | 27 | 27 | 30 | 28 | 129
  More than one race | 0 | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 2 | 1 | 10
  Not Hispanic or Latino | 14 | 28 | 26 | 28 | 29 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 29 | 28 | 30 | 30 | 135

OUTCOME MEASURES:

1. Secondary Outcome: Mean Daily Insulin Dose
Description: Prandial insulin doses were recorded during 10-point glucose monitoring for a total of 3 days during each treatment period (3 days during Week 10 of Treatment Period 1 and 3 days during Week 22 of Treatment Period 2). The mean daily insulin dose over the 3 days during each treatment period is presented. Data is presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts).
Time Frame: Week 10 and Week 22
Population: Participants who completed both Treatment Period 1 and Treatment Period 2 and had evaluable insulin dose data.
Measure: Mean (Standard Deviation); unit: units (U)
Groups:
- Analog-PH20: 100 units per milliliter (U/mL) insulin lispro or insulin aspart with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously (SC), pre-meals, for 12 weeks, with doses titrated to each participant individually
- Insulin Lispro: 100 units per milliliter (U/mL) insulin lispro, injected subcutaneously (SC), pre-meals, for 12 weeks, with doses titrated to each participant individually
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 102 | 105
units (U) | 54.28 (27.071) | 56.05 (27.243)

2. Secondary Outcome: Percentage of Participants Meeting Glucose Targets
Description: Participants were instructed to monitor their blood glucose levels a minimum of 4 times per day on all non-10-point glucose monitoring days. The number of participants meeting 90-minute postprandial plasma glucose (PPG) targets of <140 and <180 milligrams per deciliter (mg/dL) for at least 2/3 of values during non-10-point glucose monitoring days was recorded. The percentage was calculated by dividing the number of participants with values meeting the specified target at least 2/3 of the time by the total number of participants analyzed, multiplied by 100. Data is presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts).
Time Frame: Baseline through Week 24, excluding 10-point glucose monitoring days
Population: Participants who completed both Treatment Period 1 and Treatment Period 2 and had evaluable postprandial glucose data.
Measure: Number; unit: percentage of participants
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 113 | 113
percentage of participants
  PPG <140 mg/dL for all meals | 15.0 | 8.8
  PPG <140 mg/dL for breakfast: number analyzed (Participants) | 112 | 113
  PPG <140 mg/dL for breakfast | 21.4 | 10.6
  PPG <180 mg/dL for all meals | 69.9 | 59.3
  PPG <180 mg/dL for breakfast: number analyzed (Participants) | 112 | 113
  PPG <180 mg/dL for breakfast | 70.5 | 54.0

3. Secondary Outcome: Rates of Hypoglycemia at the End of Each Treatment Period
Description: Overall rates of hypoglycemia (blood glucose ≤70 milligrams per deciliter [mg/dL] and <56 mg/dL) were calculated based on 4 weeks of observation for each treatment period. Data is presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts). A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Week 12 and Week 24
Population: Participants who completed both Treatment Period 1 and Treatment Period 2.
Measure: Number; unit: events per participant per month
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 113 | 113
events per participant per month
  ≤70 mg/dL | 18.96 | 19.91
  <56 mg/dL: number analyzed (Participants) | 112 | 112
  <56 mg/dL | 7.50 | 8.05

4. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1C (HbA1c) at the End of Each Treatment Period
Description: Glycosylated hemoglobin A1C (HBA1c) levels were measured at baseline (Week 0) and at the end of each treatment period (Week 12 and Week 24). Data are presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts). Least Squares (LS) means were calculated from mixed effects linear models with treatment (Lispro, Aspart), recombinant human hyaluronidase PH20 (rHuPH20; yes, no), and treatment sequence as fixed effects and participant within treatment sequence as a random effect.
Time Frame: Baseline, Week 12 and Week 24
Population: Participants who completed both Treatment Period 1 and Treatment Period 2 and had evaluable hemoglobin A1C data.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin A1C
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 111 | 110
percentage of hemoglobin A1C | -0.14 (0.415) | -0.19 (0.440)
Statistical Analysis 1: Comparison: Analog-PH20 vs Insulin Lispro; Approximately 110 participants were to be enrolled, allowing approximately 88 participants to complete both treatment periods (44 for each investigational drug). Assuming a dropout rate of no more than 20%, intra-participant correlation of 0.80, standard deviation of 1.2, and a true difference of 0, the study would have a greater than 90% power to show that Analog-PH20 was non-inferior to insulin lispro alone with respect to the change from baseline in A1C at the end of each treatment period; Test type: Non-Inferiority or Equivalence — Non-inferiority would be supported if the upper limit of the two-sided 95% confidence interval for the difference between Analog-PH20 and the comparator (insulin lispro) did not exceed 0.40; p = 0.2878, Mixed Models Analysis; LS Means Difference = 0.05, 95% CI 2-sided [-0.05 to 0.15]

5. Secondary Outcome: Change From Baseline in Body Weight at the End of Each Treatment Period
Description: Body weight was measured at baseline (Week 0) and at the end of each treatment period (Week 12 and Week 24). Data is presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts).
Time Frame: Baseline, Week 12 and Week 24
Population: Participants who completed both Treatment Period 1 and Treatment Period 2 and had evaluable body weight data.
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 113 | 113
pounds (lbs) | -0.25 (5.702) | 0.10 (4.601)

6. Secondary Outcome: Mean Daily Postprandial Glucose (PPG) Excursions
Description: Participants performed 10-point glucose monitoring for a total of 3 days during each treatment period (3 days during Week 10 of Treatment Period 1 and 3 days during Week 22 of Treatment Period 2). Mean daily postprandial plasma glucose (PPG) excursions (referring to the change in blood glucose levels from before to after a meal) during 10-point glucose monitoring for breakfast, lunch, and dinner are presented. Data were collected 1 and 2 hours (hr) after each meal for 3 days and the means of each excursion are presented.
Time Frame: Week 10 and Week 22
Population: Participants who completed both Treatment Period 1 and Treatment Period 2 and had evaluable postprandial glucose (PPG) excursion data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 102 | 106
milligrams per deciliter (mg/dL)
  1-hr breakfast excursion: number analyzed (Participants) | 102 | 105
  1-hr breakfast excursion | 18.85 (48.348) | 27.46 (43.938)
  2-hr breakfast excursion: number analyzed (Participants) | 101 | 106
  2-hr breakfast excursion | -5.63 (52.657) | 7.08 (56.997)
  1-hr lunch excursion: number analyzed (Participants) | 100 | 104
  1-hr lunch excursion | 16.26 (46.524) | 26.25 (39.070)
  2-hr lunch excursion: number analyzed (Participants) | 101 | 104
  2-hr lunch excursion | 10.68 (53.787) | 20.77 (47.005)
  1-hr dinner excursion | -0.31 (41.368) | 4.47 (52.986)
  2-hr dinner excursion | -5.13 (46.956) | -5.16 (54.309)

ADVERSE EVENTS:
Description: Adverse event data were collected in the Intent-to-Treat (ITT) analysis set, defined as all participants who received at least one injection of study drug during a treatment period and had any efficacy endpoint data collected.
Groups:
- Titration Period (All Enrolled Participants): Prior to randomization, all enrolled participants underwent a titration period of 4-6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually.
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Lispro-PH20 Treatment Period: 100 units per milliliter (U/mL) insulin lispro with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Insulin Lispro (Lispro-PH20 Cohort) Treatment Period: Participants were randomized to the Lispro-PH20 cohort.
  100 units per milliliter (U/mL) insulin lispro, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Aspart-PH20 Treatment Period: 100 units per milliliter (U/mL) insulin aspart with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Insulin Lispro (Aspart-PH20 Cohort) Treatment Period: Participants were randomized to the Aspart-PH20 cohort.
  100 units per milliliter (U/mL) insulin lispro, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
Arm/Group | Titration Period (All Enrolled Participants) | Lispro-PH20 Treatment Period | Insulin Lispro (Lispro-PH20 Cohort) Treatment Period | Aspart-PH20 Treatment Period | Insulin Lispro (Aspart-PH20 Cohort) Treatment Period
Serious Adverse Events (participants affected / at risk) | 2/135 | 0/56 | 1/57 | 0/58 | 1/59
Other Adverse Events (participants affected / at risk) | 48/135 | 34/56 | 29/57 | 27/58 | 30/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Titration Period (All Enrolled Participants) (N=135) | Lispro-PH20 Treatment Period (N=56) | Insulin Lispro (Lispro-PH20 Cohort) Treatment Period (N=57) | Aspart-PH20 Treatment Period (N=58) | Insulin Lispro (Aspart-PH20 Cohort) Treatment Period (N=59)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Titration Period (All Enrolled Participants) (N=135) | Lispro-PH20 Treatment Period (N=56) | Insulin Lispro (Lispro-PH20 Cohort) Treatment Period (N=57) | Aspart-PH20 Treatment Period (N=58) | Insulin Lispro (Aspart-PH20 Cohort) Treatment Period (N=59)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0/61 | 0/26 | 1/26 | 0/28 | 0/29
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 2 | 2 | 3
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0/61 | 0/26 | 0/26 | 0/28 | 1/29
Headache (Nervous system disorders) | 2 | 1 | 1 | 4 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 2 | 2 | 1 | 0
Influenza like illness (General disorders) | 2 | 2 | 2 | 0 | 1
Injection site erythema (General disorders) | 1 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 1
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site urticaria (General disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 8 | 8 | 8 | 6
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 5 | 2 | 3 | 5 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Stress at work (Social circumstances) | 0 | 1 | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Trochanteric syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 3 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Weight increased (Investigations) | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.